CLINICAL TRIAL: NCT05918939
Title: Immunobridging Study: Immunogenicity and Safety of Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) Vaccine as Heterologue Booster in Adult Subjects in Indonesia
Brief Title: UNAIR Inactivated COVID-19 Vaccine as Heterologue Booster (Immunobridging Study)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Indonesia-MoH (Other Government); Universitas Airlangga (Other); Bioxis Pharmaceuticalls (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNAIR-MP-INAKTIF-BO-007
Record Dates: First submitted 2023-06-21; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pandemic; COVID-19 Vaccines
Keywords: Inactivated COVID-1 9 Vaccine; Inactivated COVID-1 9 Booster Vaccine; Immunogenicity; Safety; COVID-19; Indonesia; Immunobridging Study
MeSH Terms: conditions — COVID-19 | interventions — vaksin merah putih - UA SARS-CoV-2 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: There will be 2 groups in the study. First group will receive CoronaVac vaccine, manwhile the other group will receive Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine.
Who Masked: Participant, Investigator
Masking Description: This is an observer blind randomized controlled trial. There will be 2 groups in the trial. All subjects will have either CoronaVac or Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine as booster injection. There will be 350 subjects in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) 5 µg (Experimental): Study product are provided in the form of liquid in vial (1 ml per vial). The vaccine will be given 1 dose (0.5 ml) once.
  Interventions: Biological: Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) 5 µg
- CoronaVac Biofarma COVID-1 9 Vaccine 3 µg (Active Comparator): Control vaccine is CoronaVac Bio Farma vaccine, supplied by Ministry of Health of Indonesia, in the form of one dose vial (0.5 ml) once.
  Interventions: Biological: CoronaVac Biofarma COVID-1 9 Vaccine 3 µg

INTERVENTIONS:
Biological: Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) 5 µg — Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) contains purified S protein of SARSCoV-2 - Dose: 5 µg, aluminium hydroxide gel, 10 mM L-Histidine buffer, 0.005%, Tween Polysorbate 80, and 0.9% Sodium chloride. Vaccine will be prepared in vial
  (1 ml per vial). The vial should be shaken well before injection.
  Arms: Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) 5 µg
Biological: CoronaVac Biofarma COVID-1 9 Vaccine 3 µg — Control vaccine in this study is existing CoronaVacBioFarma inactivated COVID-19 vaccine which has been used widely in Indonesia.
  Arms: CoronaVac Biofarma COVID-1 9 Vaccine 3 µg

SUMMARY:
This is an observer blind randomized controlled trial study to evaluate the humoral immunogenicity profile - neutralizing antibody - after 28 days following vaccination with Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine as heterologue booster compared with CoronaVac administered intramuscularly in healthy adults age 18 year and above.

Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine is an inactivated vaccine made of SARS-CoV-2 virus isolated from a patient in Surabaya, composed with aluminium hydroxy gel, tween 80, and L-histidine, and this will be the first booster study in human.

DETAILED DESCRIPTION:
This is an observer blind randomized controlled trial. There will be 2 groups in the study. First group will receive CoronaVac vaccine, manwhile the other group will receive Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine. The inclusion and exclusion criteria for the subjects were listed below. All subjects will receive either one dose of CoronaVac or Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine and be followed for 6 months. The vaccine will be administered intramuscularly.

This study will have one interim and one full analysis reports. The main focus is immunogenicity and safety issues.

Data Safety Monitoring Board will be commissioned for this study to evaluate safety data over the study period and to review any events that meet a specific study pausing rule or any other safety issue that may arise. They will review the blinded 7 and 28 days safety data following the vaccine, and then the 3 and 6 months safety data. The immunogenicity data will be evaluated until 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults and elderly, males and females, 18 years of age and above. Healthy status will be determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
2. Subjects already received 2 (two) doses of CoronaVac inactivated vaccines at least 6 months prior to this study.
3. Subjects have been informed properly regarding the study and signed the informed consent form
4. Subject will commit to comply with the instructions of the investigator and the schedule of the trial
5. Female subjects of childbearing potential must agree to consistently use any methods of contraception (except the periodic abstinence) from at least 21 days prior to enrollment and through 6 months after the vaccination.
6. Participants agree not to donate bone marrow, blood, and blood products from the vaccine administration until 3 months after receiving the vaccine.
7. Participants must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another vaccine trial
2. Evolving mild, moderate, and severe illness, especially infectious diseases or fever (axillary temperature 37.5oC or more) concurrent or within 7 days prior to study vaccination. This includes respiratory or constitutional symptms consistent with SARS-CoV-2 (cough, sore throat, difficulty in breathing, etc)
3. Known history of allergy to any component of the vaccines
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
5. Any autoimmune or immunodeficiency disease/condition
6. Subjects who have received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood derived products, long term corticosteroid - more than 2 weeks, and so on), OR anticipation of the need for immunosuppressive treatment within 6 months after last vaccination. The use of topical or nasal steroid will be permitted. Inhaled glucocorticoids are prohibited.
7. Unstable chronic disease, inclusive of uncontrolled hypertension, congestive heart failure, chronic obstructive pulmonary disease, asthma, chronic urticaria, diabetes requiring use of medicine. The final decision regarding this condition will be decided by the attending field clinicians or investigator.
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
9. Individuals who previously receive any booster vaccine against Covid-19.
10. Individuals who have a previously ascertained Covid-19 in the period of 1 month (for mild, moderate, or asymptomatic people) or 3 months (for severe Covid-19) before the recruit of this study, or in a close contact in the last 14 days with confirmed case of Covid-19.
11. Positive test for SARS-CoV-2 (Antigen or PCR) at screening prior to the vaccination. Testing may be repeated during the screening period if exposure to positive confirmed case of SARS-CoV-2 is suspected, at the discretion of investigator.
12. History of alcohol or substance abuse
13. HIV patients.
14. Malignancy patients within 3 years prior to study vaccination.
15. Any neurological disease or history of significant neurological disorder such as meningitis, encephalitis, Guillain-Barre Syndrome, multiple sclerosis, etc
16. Vital sign abnormalities and clinical laboratory abnormalities as decided by the investigators. Vital sign measurements and clinical laboratory testing may be repeated before the final decision.
17. Women who are pregnant or who plan to become pregnant during the study.
18. Participant has major psychiatric problem or illness
19. Participant cannot communicate reliably with the investigator
20. Participant has contraindication to intramuscular injection and blood draws, such as bleeding disorders or phobia.
21. Participant had major surgery within 12 weeks before vaccination which will not be fully recovered, or has major surgery planned during the time participant is expected to participate in the study or within 6 months after the last dose of study vaccine administration.
22. Any condition that in the opinion of the investigators would pose a helath risk to the subject if enrolled or could interfere with the evaluation of the vaccine or interpretation of the study results
23. Study team members.
24. Subject planning to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-08-05 (Estimated); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
The Humoral Immunogenicity Profile | 28 days after the booster vaccination
  The level of neutralizing antibody - after 28 days following vaccination with Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine as heterologue booster compared with CoronaVac administered intramuscularly in healthy adults age 18 year and above

OTHER OUTCOMES:
Safety and reactogenicity | Within 7 and 28 days, 3 and 6 months following vaccination
  Evaluate number of adverse events occur among participants
The Humoral Immune Response - Neutralizing Antibody | 3 and 6 months following the booster vaccination
  The level of neutralizing antibody after 3 and 6 months following vacciation with Vaksin Merah Putih - UA SARS-CoV-2 (Vero Cell Inactivated) vaccine as heterologue booster compared with CoronaVac administered intramuscularly in healthy adults age 18 year and above.
The Humoral Immune Response - Non Neutralizing Antibody | at 28 days, 3 and 6 months following vaccination
  The level of non neutralizing titers in serum following vaccination with Vaksin Merah Putih - UA SARSCoV-2 (Vero Cell Inactivated) vaccine as heterologue booster compared with CoronaVac administered intramuscularly in healthy adults age 18 year and above

CONTACTS AND LOCATIONS:
Overall Officials: Dominicus Husada, MD, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Wang Z, Wang G, Lau JY, Zhang K, Li W. COVID-19 in early 2021: current status and looking forward. Signal Transduct Target Ther. 2021 Mar 8;6(1):114. doi: 10.1038/s41392-021-00527-1. PMID 33686059
- [Background] Noh JY, Song JY, Yoon JG, Seong H, Cheong HJ, Kim WJ. Safe hospital preparedness in the era of COVID-19: The Swiss cheese model. Int J Infect Dis. 2020 Sep;98:294-296. doi: 10.1016/j.ijid.2020.06.094. Epub 2020 Jun 30. PMID 32619759
- [Background] New York Vaccine Tracker. Downloaded from https://www.nytimes.com/interactive/2020/science/coronavirus-vaccinetracker.html. Accessed 30 April 2022.
- [Background] Badan POM Republik Indonesia. Dowloaded from https://www.pom.go.id/new/view/more/pers/605/Pastikan-Keamanan-danMutu-Vaksin---Badan-POM-Kawal-Uji-Klinik-Vaksin-Merah-Putih.html. Accessed 11 October 2021.
- [Background] Irwin A. What it will take to vaccinate the world against COVID-19. Nature. 2021 Apr;592(7853):176-178. doi: 10.1038/d41586-021-00727-3. No abstract available. PMID 33767468
- [Background] So AD, Woo J. Reserving coronavirus disease 2019 vaccines for global access: cross sectional analysis. BMJ. 2020 Dec 15;371:m4750. doi: 10.1136/bmj.m4750. PMID 33323376
- [Background] Worldometer coronavirus cases. Downloaded from https://www.worldometers.info/coronavirus/. Accessed 30 April 2022.
- [Background] Biswas M, Rahaman S, Biswas TK, Haque Z, Ibrahim B. Association of Sex, Age, and Comorbidities with Mortality in COVID-19 Patients: A Systematic Review and Meta-Analysis. Intervirology. 2020 Dec 9:1-12. doi: 10.1159/000512592. Online ahead of print. PMID 33296901
- [Background] Satuan Tugas Penanganan Covid-19. Downloaded from https://covid19.go.id/petasebaran. Accessed 30 April 2022.
- [Background] Cirrincione L, Plescia F, Ledda C, Rapisarda V, Martorana D, Moldovan RE, Theodoridou K, Cannizzaro E. COVID-19 Pandemic: Prevention and Protection Measures to Be Adopted at the Workplace. Sustainability 2020; 12: 3603.
- [Background] Bloomberg. Downloaded from https://www.bloomberg.com/graphics/covidresilience-ranking/. Accessed 11 October 2021.
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Background] Our world in Data. Downloaded from https://ourworldindata.org/covid-vaccinations. Accessed 30 April 2022.
- [Background] CNN. Downloaded from https://edition.cnn.com/2021/04/03/health/us-coronavirussaturday/index.html. Accessed 11 October 2021.
- [Background] World Health Organization. Downloaded from https://www.who.int/newsroom/feature-stories/detail/vaccine-efficacy-effectiveness-and-protection. Accessed 11 October 2021.
- [Background] Palacios R, Patino EG, de Oliveira Piorelli R, Conde MTRP, Batista AP, Zeng G, Xin Q, Kallas EG, Flores J, Ockenhouse CF, Gast C. Double-Blind, Randomized, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of treating Healthcare Professionals with the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac - PROFISCOV: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 15;21(1):853. doi: 10.1186/s13063-020-04775-4. PMID 33059771
- [Background] Tanriover MD, Doganay HL, Akova M, Guner HR, Azap A, Akhan S, Kose S, Erdinc FS, Akalin EH, Tabak OF, Pullukcu H, Batum O, Simsek Yavuz S, Turhan O, Yildirmak MT, Koksal I, Tasova Y, Korten V, Yilmaz G, Celen MK, Altin S, Celik I, Bayindir Y, Karaoglan I, Yilmaz A, Ozkul A, Gur H, Unal S; CoronaVac Study Group. Efficacy and safety of an inactivated whole-virion SARS-CoV-2 vaccine (CoronaVac): interim results of a double-blind, randomised, placebo-controlled, phase 3 trial in Turkey. Lancet. 2021 Jul 17;398(10296):213-222. doi: 10.1016/S0140-6736(21)01429-X. Epub 2021 Jul 8. PMID 34246358
- [Background] Reuters. Downloaded from https://www.reuters.com/business/healthcarepharmaceuticals/indonesia-study-finds-chinas-sinovac-covid-19-vaccine-effectivemedical-staff-2021-05-12/. Accessed 11 October 2021.
- [Background] Al Kaabi N, Zhang Y, Xia S, Yang Y, Al Qahtani MM, Abdulrazzaq N, Al Nusair M, Hassany M, Jawad JS, Abdalla J, Hussein SE, Al Mazrouei SK, Al Karam M, Li X, Yang X, Wang W, Lai B, Chen W, Huang S, Wang Q, Yang T, Liu Y, Ma R, Hussain ZM, Khan T, Saifuddin Fasihuddin M, You W, Xie Z, Zhao Y, Jiang Z, Zhao G, Zhang Y, Mahmoud S, ElTantawy I, Xiao P, Koshy A, Zaher WA, Wang H, Duan K, Pan A, Yang X. Effect of 2 Inactivated SARS-CoV-2 Vaccines on Symptomatic COVID-19 Infection in Adults: A Randomized Clinical Trial. JAMA. 2021 Jul 6;326(1):35-45. doi: 10.1001/jama.2021.8565. PMID 34037666
- [Background] Kyriakidis NC, Lopez-Cortes A, Gonzalez EV, Grimaldos AB, Prado EO. SARS-CoV-2 vaccines strategies: a comprehensive review of phase 3 candidates. NPJ Vaccines. 2021 Feb 22;6(1):28. doi: 10.1038/s41541-021-00292-w. PMID 33619260
- [Background] Mendonca SA, Lorincz R, Boucher P, Curiel DT. Adenoviral vector vaccine platforms in the SARS-CoV-2 pandemic. NPJ Vaccines. 2021 Aug 5;6(1):97. doi: 10.1038/s41541-021-00356-x. PMID 34354082
- [Background] Yadav T, Srivastava N, Mishra G, Dhama K, Kumar S, Puri B, Saxena SK. Recombinant vaccines for COVID-19. Hum Vaccin Immunother. 2020 Dec 1;16(12):2905-2912. doi: 10.1080/21645515.2020.1820808. Epub 2020 Nov 24. PMID 33232211
- [Background] Badan POM Republik Indonesia. Downloaded from https://www.pom.go.id/new/view/more/pers/629/Badan-POM-Terbitkan-EUAVaksin-Covovax-Sebagai-Vaksin-Alternatif-Ke-11-dalam-Penanganan-Pandemi.html. Accessed 11 April 2022.
- [Background] Pollard AJ, Bijker EM. A guide to vaccinology: from basic principles to new developments. Nat Rev Immunol. 2021 Feb;21(2):83-100. doi: 10.1038/s41577-020-00479-7. Epub 2020 Dec 22. PMID 33353987
- [Background] Excler JL, Saville M, Berkley S, Kim JH. Vaccine development for emerging infectious diseases. Nat Med. 2021 Apr;27(4):591-600. doi: 10.1038/s41591-021-01301-0. Epub 2021 Apr 12. PMID 33846611
- [Background] Bhattacharya S, Dasgupta R. Smallpox and polio eradication in India: comparative histories and lessons for contemporary policy. Cien Saude Colet. 2011 Feb;16(2):433-44. doi: 10.1590/s1413-81232011000200007. PMID 21340319
- [Background] Jayk Bernal A, Gomes da Silva MM, Musungaie DB, Kovalchuk E, Gonzalez A, Delos Reyes V, Martin-Quiros A, Caraco Y, Williams-Diaz A, Brown ML, Du J, Pedley A, Assaid C, Strizki J, Grobler JA, Shamsuddin HH, Tipping R, Wan H, Paschke A, Butterton JR, Johnson MG, De Anda C; MOVe-OUT Study Group. Molnupiravir for Oral Treatment of Covid-19 in Nonhospitalized Patients. N Engl J Med. 2022 Feb 10;386(6):509-520. doi: 10.1056/NEJMoa2116044. Epub 2021 Dec 16. PMID 34914868
- [Background] Mahase E. Covid-19: Pfizer's paxlovid is 89% effective in patients at risk of serious illness, company reports. BMJ. 2021 Nov 8;375:n2713. doi: 10.1136/bmj.n2713. No abstract available. PMID 34750163
- [Background] CNN Indonesia. Downloaded from https://www.cnnindonesia.com/ekonomi/20210615172504-92-654688/bio-farmayakin-ri-bisa-dapat-400-juta-dosis-vaksin-tahun-ini. Accessed 11 October 2021.
- [Background] Suara.com. Downloaded from https://www.suara.com/bisnis/2020/11/06/151502/ini-6-lembaga-yangkembangkan-vaksin-merah-putih. Accessed 11 October 2021.
- [Background] Abbasi J. Studies Suggest COVID-19 Vaccine Boosters Save Lives. JAMA. 2022 Jan 11;327(2):115. doi: 10.1001/jama.2021.23455. No abstract available. PMID 35015054
- [Background] Burckhardt RM, Dennehy JJ, Poon LLM, Saif LJ, Enquist LW. Are COVID-19 Vaccine Boosters Needed? The Science behind Boosters. J Virol. 2022 Feb 9;96(3):e0197321. doi: 10.1128/JVI.01973-21. Epub 2021 Nov 24. PMID 34817198
- [Background] Mattiuzzi C, Lippi G. Efficacy of COVID-19 vaccine booster doses in older people. Eur Geriatr Med. 2022 Feb;13(1):275-278. doi: 10.1007/s41999-022-00615-7. Epub 2022 Jan 24. PMID 35067909
- [Background] Parker EPK, Desai S, Marti M, Nohynek H, Kaslow DC, Kochhar S, O'Brien KL, Hombach J, Wilder-Smith A. Response to additional COVID-19 vaccine doses in people who are immunocompromised: a rapid review. Lancet Glob Health. 2022 Mar;10(3):e326-e328. doi: 10.1016/S2214-109X(21)00593-3. No abstract available. PMID 35180408